CLINICAL TRIAL: NCT00002519
Title: PH I Continuous Infusion Taxol in Combination With Thoracic Radiation Therapy in Untreated Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Paclitaxel Plus Radiation Therapy in Treating Patients With Untreated Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: David Carbone, M.D., Ph.D., Vanderbilt-Ingram Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VCC LUN65; P30CA068485 (NIH); VU-VCC-LUN-65; UPCC-3597; NCI-T92-0246D
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy with paclitaxel in combination with radiation therapy to the chest in patients with previously untreated stage III non-small cell lung cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of paclitaxel when combined with standard thoracic radiotherapy in patients with locally advanced non-small cell lung cancer. II. Determine the plasma levels of paclitaxel in these patients. III. Determine the effect of this regimen on the tumor cell cycle distribution in these patients.

OUTLINE: This is a dose-escalation study of paclitaxel. Patients undergo standard thoracic radiotherapy 5 days a week for 7 weeks. Patients receive paclitaxel IV continuously beginning 48 hours before initiating radiotherapy and continuing until the last day of radiotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-5 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 5 patients experience dose-limiting toxicity. Patients are followed monthly for 2 years.

PROJECTED ACCRUAL: A total of 3-5 patients per dose level will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven previously untreated non-small cell lung cancer that is not amenable to potentially curative surgery due to the following: Direct invasion of the mediastinum, heart, great vessels, trachea, esophagus, vertebral body, or carina by tumor (T4) Cytologically positive scalene or supraclavicular nodes Mediastinal or contralateral hilar nodes 3 cm or greater on CT, with or without pathological confirmation Pathologically positive mediastinal or contralateral hilar nodes on mediastinoscopy or Chamberlain procedure (N2 or N3) Medically inoperable stage IIIA disease (e.g., resection would result in insufficient pulmonary volume) allowed No distant metastases No pleural effusion (regardless of fluid cytology) Evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 0-2 Hematopoietic: WBC normal Platelet count normal Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) Transaminases no greater than 2 times ULN Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No significant coronary artery disease No documented myocardial infarction No angina, arrhythmia, or congestive heart failure requiring medication Pulmonary: FEV1 greater than 1 liter pO2 greater than 55 mm Hg on room air pCO2 less than 45 mm Hg on room air Other: No prior severe hypersensitivity reaction to products containing Cremaphor EL No clinical evidence of pre-existing polyneuropathy Not pregnant Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior thoracic irradiation Surgery: See Disease Characteristics Other: No concurrent medications known to alter cardiac conduction or cause bradycardia (e.g., digoxin, beta blockers, or calcium channel blockers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1997-01; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Carbone, MD, PhD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee